CLINICAL TRIAL: NCT06199102
Title: The High Initial Dose of Monitored Vitamin D Supplementation in Preterm Infants. A Randomized Controlled Study.
Brief Title: The High Initial Dose of Monitored Vitamin D Supplementation in Preterm Infants.
Acronym: HIDVID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Alicja Kołodziejczyk, MD, PhD, Princess Anna Mazowiecka Hospital, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VitD-2023
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Vitamin D Deficiency; Osteopenia of Prematurity; Nephrolithiasis; Metabolic Bone Disease; Late-Onset Neonatal Sepsis
Keywords: vitamin D; preterm infants; osteopenia of prematurity; late-onset sepsis; metabolic bone disease
MeSH Terms: conditions — Vitamin D Deficiency; Bone Diseases, Metabolic; Nephrolithiasis; Neonatal Sepsis | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monitored group (Experimental): Infants in the monitored group will receive an initial dose of 1000 IU of vit D (cholecalciferol/ Devikap; Polpharma, Starogard Gdański, Poland).
  Interventions: Dietary Supplement: cholecalciferol/ Devikap
- controlled group (Active Comparator): Infants in the controlled group will receive 250 IU (cholecalciferol/ Devikap; Polpharma, Starogard Gdański, Poland) for very low birth weight infants and 500 IU (cholecalciferol/ Devikap; Polpharma, Starogard Gdański, Poland) for infants weighing above 1000 g.
  Interventions: Dietary Supplement: cholecalciferol/ Devikap

INTERVENTIONS:
Dietary Supplement: cholecalciferol/ Devikap — Infants in the monitored group will receive an initial dose of 1000 IU of vit D. An additional 160 IU/kg of vit D is included in parenteral nutrition, as well as 150-300 IU/kg in enteral nutrition, depending on the amount and source of enteral feeding (i.e., human milk fortifiers or milk formula). At 28±2 days of age, blood samples will be obtained for 25(OH)D concentration measurement, followed by measurements every 4 weeks and/or 35±1 weeks of PCA. In the monitored group, vit D doses will be appropriately modified, based on 25(OH)D levels, using the scheme described in the Polish recommendation. The intake from the diet will be calculated from the second month of life.
  Arms: monitored group
Dietary Supplement: cholecalciferol/ Devikap — Infants in the controlled group will receive 250 IU for very low birth weight infants and 500 IU for infants weighing above 1000 g. An additional 160 IU/kg of vit D is included in parenteral nutrition, as well as 150-300 IU/kg in enteral nutrition, depending on the amount and source of enteral feeding (i.e., human milk fortifiers or milk formula). Infants assigned to the standard therapy group will undergo the same blood sample collection procedure as the monitored group, but without any alterations in their dosing regimen.
  Arms: controlled group

SUMMARY:
The aim of this study will be to assess the effectiveness of monitored vit D supplementation in a population of preterm infants and to identify whether the proper vit D supplementation in preterm infants can reduce the incidence of neonatal sepsis and incidence of metabolic bone disease.

DETAILED DESCRIPTION:
Vitamin D deficiency can escalate prematurity bone disease in preterm infants and negatively influence their immature immunology system. Infants born at 24+0/7 weeks to 32+6/7 weeks of gestation will be considered for inclusion. Cord or vein blood samples will be obtained within 48 h after birth for 25-hydroxyvitamin D level measurements. Parathyroid hormone and interleukin-6 levels will be measured. Infants will be randomized to the monitored group (i.e., initial dose of 1000 IU/day and possible modification) or the controlled group (i.e., 250 IU/day or 500 IU/day dose, depending on weight). Supplementation will be monitored up to postconceptional age 35 weeks. The primary endpoint is the percentage of infants with deficient or suboptimal 25-hydroxyvitamin D levels at 28±2 days of age. 25-Hydroxyvitamin D levels will be measured at postconceptional age 35±2 weeks. Secondary objectives include the incidence of sepsis, osteopenia, hyperparathyroidism, and elevated interleukin-6 concentration. The aim of this study will be to assess the effectiveness of monitored vitamin D supplementation in a population of preterm infants and to determine whether a high initial dose of monitored vitamin D supplementation in preterm infants can reduce the incidence of neonatal sepsis and incidence of metabolic bone disease.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with a gestational age of 24+0/7 to 32+6/7 born at our clinic
* preterm infants with a gestational age of 24+0/7 to 32+6/7 outborn and admitted to our intensive care unit within 48h after delivery
* written informed consent form caregivers for the mother and the child to participate in the study

Exclusion Criteria:

* infants born at >32 weeks of gestation
* infants with major congenital abnormalities or other severe congenital malformations
* infants with genetic disorders (diagnosed before and after birth) deemed incompatible with survival
* infants with diagnosed cholestasis
* the absence of written informed consent and challenges in communication with caregivers

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of infants with deficient or suboptimal 25(OH)D levels. | at 28±2 days of age, after that every 4 weeks (number of measurements depends on gestation age at birth) and/ or at 35±1 weeks of postconceptional age
  25-hydroxyvitamin D serum level below 30ng/ml

SECONDARY OUTCOMES:
The number of infants with neonatal late-onset sepsis. | after 3 days of age
  blood culture-proven (one blood sample of at least 1 mL) and/or clinical sepsis occurring after 3 days of age
The number of infants with biochemical markers of metabolic bone disease. | at 35±1 weeks of postconceptional age
  serum levels of alkaline phosphatase >500 IU and serum phosphate <1.8 mmol/L
The number of infants with hyperparathyroidism. | at birth, at 28±2 days of life, and at 35±1 weeks of postconceptional age
  serum or plasma concentration of PTH in infants should be 10-40 pg/mL
The number of infants with high interleukin-6 levels. | at birth, at 28±2 days of life, and at 35±1 weeks of postconceptional age
  the reference interval is calculated as 44 pg/mL; it is released within 2 h after the onset of bacteremia, peaks at approximately 6 h, and finally declines over the following 24 h
The number of infants with nephrocalcinosis and nephrolithiasis. | at 28±2 days of life and at 35±1 weeks of postconceptional age
  venous samples for serum and urine calcium, and creatinine level measurements
The number of infants with potentially toxic 25(OH)D levels. | at 28±2 days of age, after that every 4 weeks (number of measurements depends on gestation age at birth) and/ or at 35±1 weeks of postconceptional age
  25-hydroxyvitamin D serum level exceeding 100 ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Renata Bokiniec, MD, PhD, Study Chair — renata.bokiniec@wum.edu.pl
Locations (1):
- Princess Anna Mazowiecka Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lips P, van Schoor NM. The effect of vitamin D on bone and osteoporosis. Best Pract Res Clin Endocrinol Metab. 2011 Aug;25(4):585-91. doi: 10.1016/j.beem.2011.05.002. PMID 21872800
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Shaker JL, Deftos L. Calcium and Phosphate Homeostasis. 2023 May 17. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK279023/ PMID 25905252
- [Background] Khundmiri SJ, Murray RD, Lederer E. PTH and Vitamin D. Compr Physiol. 2016 Mar 15;6(2):561-601. doi: 10.1002/cphy.c140071. PMID 27065162
- [Background] Thorsen SU, Pipper CB, Skogstrand K, Pociot F, Svensson J. 25-Hydroxyvitamin D and Peripheral Immune Mediators: Results from Two Nationwide Danish Pediatric Cohorts. Nutrients. 2017 Apr 6;9(4):365. doi: 10.3390/nu9040365. PMID 28383493
- [Background] Pinto MRC, Machado MMT, de Azevedo DV, Correia LL, Leite AJM, Rocha HAL. Osteopenia of prematurity and associated nutritional factors: case-control study. BMC Pediatr. 2022 Sep 1;22(1):519. doi: 10.1186/s12887-022-03581-y. PMID 36050673
- [Background] Pludowski P, Kos-Kudla B, Walczak M, Fal A, Zozulinska-Ziolkiewicz D, Sieroszewski P, Peregud-Pogorzelski J, Lauterbach R, Targowski T, Lewinski A, Spaczynski R, Wielgos M, Pinkas J, Jackowska T, Helwich E, Mazur A, Ruchala M, Zygmunt A, Szalecki M, Bossowski A, Czech-Kowalska J, Wojcik M, Pyrzak B, Zmijewski MA, Abramowicz P, Konstantynowicz J, Marcinowska-Suchowierska E, Bleizgys A, Karras SN, Grant WB, Carlberg C, Pilz S, Holick MF, Misiorowski W. Guidelines for Preventing and Treating Vitamin D Deficiency: A 2023 Update in Poland. Nutrients. 2023 Jan 30;15(3):695. doi: 10.3390/nu15030695. PMID 36771403
- [Background] Taylor SN, Wagner CL, Hollis BW. Vitamin D supplementation during lactation to support infant and mother. J Am Coll Nutr. 2008 Dec;27(6):690-701. doi: 10.1080/07315724.2008.10719746. PMID 19155428
- [Background] Rigo J, De Curtis M, Pieltain C, Picaud JC, Salle BL, Senterre J. Bone mineral metabolism in the micropremie. Clin Perinatol. 2000 Mar;27(1):147-70. doi: 10.1016/s0095-5108(05)70011-7. PMID 10690569
- [Background] Abrams SA; Committee on Nutrition. Calcium and vitamin d requirements of enterally fed preterm infants. Pediatrics. 2013 May;131(5):e1676-83. doi: 10.1542/peds.2013-0420. Epub 2013 Apr 29. PMID 23629620
- [Background] Embleton ND, Jennifer Moltu S, Lapillonne A, van den Akker CHP, Carnielli V, Fusch C, Gerasimidis K, van Goudoever JB, Haiden N, Iacobelli S, Johnson MJ, Meyer S, Mihatsch W, de Pipaon MS, Rigo J, Zachariassen G, Bronsky J, Indrio F, Koglmeier J, de Koning B, Norsa L, Verduci E, Domellof M. Enteral Nutrition in Preterm Infants (2022): A Position Paper From the ESPGHAN Committee on Nutrition and Invited Experts. J Pediatr Gastroenterol Nutr. 2023 Feb 1;76(2):248-268. doi: 10.1097/MPG.0000000000003642. Epub 2022 Oct 28. PMID 36705703
- [Background] Kolodziejczyk-Nowotarska A, Bokiniec R, Seliga-Siwecka J. Monitored Supplementation of Vitamin D in Preterm Infants: A Randomized Controlled Trial. Nutrients. 2021 Sep 28;13(10):3442. doi: 10.3390/nu13103442. PMID 34684442
- [Background] Walker VP, Modlin RL. The vitamin D connection to pediatric infections and immune function. Pediatr Res. 2009 May;65(5 Pt 2):106R-113R. doi: 10.1203/PDR.0b013e31819dba91. PMID 19190532
- [Background] Dong Y, Speer CP. Late-onset neonatal sepsis: recent developments. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F257-63. doi: 10.1136/archdischild-2014-306213. Epub 2014 Nov 25. PMID 25425653
- [Background] Aranow C. Vitamin D and the immune system. J Investig Med. 2011 Aug;59(6):881-6. doi: 10.2310/JIM.0b013e31821b8755. PMID 21527855
- [Background] Workneh Bitew Z, Worku T, Alemu A. Effects of vitamin D on neonatal sepsis: A systematic review and meta-analysis. Food Sci Nutr. 2020 Nov 10;9(1):375-388. doi: 10.1002/fsn3.2003. eCollection 2021 Jan. PMID 33473300
- [Background] Haque KN. Definitions of bloodstream infection in the newborn. Pediatr Crit Care Med. 2005 May;6(3 Suppl):S45-9. doi: 10.1097/01.PCC.0000161946.73305.0A. PMID 15857558
- [Background] Bohnhorst B, Lange M, Bartels DB, Bejo L, Hoy L, Peter C. Procalcitonin and valuable clinical symptoms in the early detection of neonatal late-onset bacterial infection. Acta Paediatr. 2012 Jan;101(1):19-25. doi: 10.1111/j.1651-2227.2011.02438.x. Epub 2011 Aug 29. PMID 21824193
- [Background] Mercy J, Dillon B, Morris J, Emmerson AJ, Mughal MZ. Relationship of tibial speed of sound and lower limb length to nutrient intake in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2007 Sep;92(5):F381-5. doi: 10.1136/adc.2006.105742. Epub 2007 Mar 16. PMID 17369280
- [Background] Rustico SE, Calabria AC, Garber SJ. Metabolic bone disease of prematurity. J Clin Transl Endocrinol. 2014 Jul 4;1(3):85-91. doi: 10.1016/j.jcte.2014.06.004. eCollection 2014 Sep. PMID 29159088
- [Background] Shahkar L, Keshtkar A, Mirfazeli A, Ahani A, Roshandel G. The role of IL-6 for predicting neonatal sepsis: a systematic review and meta-analysis. Iran J Pediatr. 2011 Dec;21(4):411-7. PMID 23056824
- [Background] Eichberger J, Resch B. Reliability of Interleukin-6 Alone and in Combination for Diagnosis of Early Onset Neonatal Sepsis: Systematic Review. Front Pediatr. 2022 Mar 23;10:840778. doi: 10.3389/fped.2022.840778. eCollection 2022. PMID 35402358
- [Background] Prinsen JH, Baranski E, Posch H, Tober K, Gerstmeyer A. Interleukin-6 as diagnostic marker for neonatal sepsis: determination of Access IL-6 cutoff for newborns. Clin Lab. 2008;54(5-6):179-83. PMID 18780664
- [Background] Barrueto F Jr, Wang-Flores HH, Howland MA, Hoffman RS, Nelson LS. Acute vitamin D intoxication in a child. Pediatrics. 2005 Sep;116(3):e453-6. doi: 10.1542/peds.2004-2580. PMID 16140692
- [Background] Al-Kandari A, Sadeq H, Alfattal R, AlRashid M, Alsaeid M. Vitamin D Intoxication and Nephrocalcinosis in a Young Breastfed Infant. Case Rep Endocrinol. 2021 Jul 30;2021:3286274. doi: 10.1155/2021/3286274. eCollection 2021. PMID 34373793
- [Background] Staub E, Wiedmer N, Staub LP, Nelle M, von Vigier RO. Monitoring of urinary calcium and phosphorus excretion in preterm infants: comparison of 2 methods. J Pediatr Gastroenterol Nutr. 2014 Apr;58(4):404-8. doi: 10.1097/MPG.0000000000000244. PMID 24253368